CLINICAL TRIAL: NCT06712797
Title: Physical Activity and Nutrition to Halt Elevated Risk in the Pancreas Interception Center (PANTHER-PIC)
Brief Title: Physical Activity and Nutrition to Halt Elevated Risk in the Pancreas Interception Center
Acronym: PANTHER-PIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Miles for Moffitt (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-23462
Record Dates: First submitted 2024-11-27; First posted 2024-12-02 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Intraductal Papillary Mucinous Neoplasm
Keywords: Pancreatic Ductal Adenocarcinoma; Intraductal Papillary Mucinous Neoplasm; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Exercise; Nutritional Status

STUDY DESIGN:
Intervention Model Description: A single-arm trial evaluating the feasibility and acceptability of a 6-month Physical Activity (PA) and Nutrition (N) intervention for Intraductal Papillary Mucinous Neoplasm (IPMN) patients who are overweight and viscerally obese (on MRI) and/or have elevated levels of SOC incretin, cytokine, or adipokine biomarkers.
  Patients with IPMNs (>15 mm) who have received or will receive care in Moffitt Cancer Center's Pancreas Interception Center (PIC) will be recruited.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity (PA) and Nutrition (N) (Experimental): Physical Activity: Participants will perform 150 minutes/week of moderate to vigorous Physical Activity per week. Participants will self-monitor physical activity using "active minutes" that approximate moderate to vigorous physical activity via a Fitbit device.
  Nutrition: Participants will undergo counseling appointments to address nutritional symptoms and will be given targets for daily calorie and protein intake following a Mediterranean diet.
  Interventions: Behavioral: Physical Activity (PA); Behavioral: Nutrition (N)

INTERVENTIONS:
Behavioral: Physical Activity (PA) — Participants will receive a Fitbit (Inspire 3, Google LLC, Mountain View, CA, USA) to encourage and self-monitor Physical Activity (PA) using "active minutes," which approximate moderate-to-vigorous PA.
  Fitbits will be synced to a HIPAA-compliant platform created by Moffitt's Biostatistics and Bioinformatics Shared Resource (BBSR).
  Study personnel will view active minutes to provide individualized feedback and encourage progression. Weekly feedback will encourage participants to increase active minutes by 10% until achieving ≥ 150 minutes to meet cancer prevention recommendations.
  Participants who reach ≥ 150 active minutes will be encouraged to maintain or exceed recommendations.
Behavioral: Nutrition (N) — Participants will undergo counseling at baseline (T0) to address nutritional symptoms and provide targets for daily calories and protein following a Mediterranean diet. This diet includes a high intake of vegetables, legumes, fruits, and unsaturated fatty acids, low intake of saturated fatty acids, and a moderately high intake of fish.
  Total caloric intake will be calculated. A standard breakdown of 40% carbohydrates, 30% fats and 30% protein will be used. Individuals will review this calculation during their office encounters and follow these values using the FitBit, application, which will adjust to their daily energy expenditure.
  Additional counseling (in-person or via Zoom) will occur at baseline (T0) + 12 weeks to gauge progress toward calorie and protein targets, monitor weight change, and guide dietary changes.
  Participants will log daily food intake and self-monitor progress toward calorie and protein goals.

SUMMARY:
The purpose of this Study is to assist in implementing a practical, easy-to-adopt lifestyle intervention that optimizes patient outcomes and minimizes pancreatic ductal adenocarcinoma (PDAC) risk.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Endoscopically, radiologically, or biopsy-proven pancreatic intraductal papillary mucinous neoplasm (IPMN) over 15 mm in size
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Ability to sign informed consent
* Ability to read and speak English or Spanish
* Body Mass Index (BMI) greater than or equal to 25 kg/m2
* Visceral obesity based on MRI quantification of visceral and subcutaneous fat; ratio of visceral to subcutaneous fat area greater than 0.4 and/or elevated cytokine, incretin or adipokine biomarkers

Exclusion Criteria:

* No diagnosis of an IPMN
* IPMN with high grade dysplasia, cancer or other high-risk features
* Screen failure for exercise safety
* Underlying unstable cardiac or pulmonary disease or symptomatic cardiac disease
* Recent fracture or acute musculoskeletal injury
* Numeric pain rating scale of 7 or more out of 10
* Myopathic or rheumatologic disease that impacts physical function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Retention Feasibility | Up to 6 Months
  Retention feasibility will be measured based on the percentage of enrolled participants who complete study assessments during the 6-month duration of enrollment (baseline T0 through follow-up T1) Target: ≥70%).
Physical Activity (PA) Adherence Feasibility | Up to 6 Months
  Adherence to Physical Activity (PA) will be based on achievement of activity minute goals (≥ 150 minutes).
  Target: 70% of participants achieve activity minute goals in ≥75% of full weeks between baseline through follow-up (T0-T1).
Nutrition (N) Adherence Feasibility | Up to 6 Months
  Adherence to Nutrition (N) will be based on completion of counseling appointments (target: 70% of participants complete both appointments) and diet logging.
  Target: 70% of participants log diet on ≥ 50% of days between baseline through follow-up (T0-T1)
Acceptability of Lifestyle Modifications | Up to 6 Months
  Acceptability will be assessed at T1 with the Participant Evaluation of Feasibility and Acceptability questionnaire, adapted to fit intervention conditions used in this study.
  This questionnaire includes Likert Scale and open-ended questions assessing difficulty and appropriateness of the Physical Acitivity (PA) and Nutrition (N) intervention components, perceived benefits, interactions with study personnel, study materials, and baseline/follow-up testing. Acceptability will be assessed on an item-by-item basis and as average item score, with scores ≥4 ("agree" to "strongly agree") indicating acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Permuth, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://www.moffitt.org/clinical-trials-research/clinical-trials/